CLINICAL TRIAL: NCT04012424
Title: The Effect of Premedication With Curcumin on Post-Operative Pain in Single Visit Endodontic Treatment of Acute Pulpitis in Mandibular Molars: A Randomized Controlled Trial
Brief Title: The Effect of Premedication With Curcumin on Post-endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Sobhy, master candidate at endodontic department faculty of dentistry cario university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 3-7-1
Record Dates: First submitted 2019-06-30; First posted 2019-07-09 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Acute Pulpitis
Keywords: curcumin as premedication - root canal treatment
MeSH Terms: interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug (400mg Curcumin) Curcumin is apice (Experimental): Curcumin is an ancient coloring spice of Asia which is powerful antioxidant , it has hepatoprotective effect and traditionally used for many remedies . Interestingly, it has various pharmacological activities including analgesic, anti-inflammatory , It is even reported to have antimicrobial effect .
  Medical clinical trials reported on the analgesic effect of curcuminoids in reducing postsurgical pain osteoarthritis and rheumatoid arthritis .
  patients will take 400mg capsule curcumin one hour before endodontic treatment and study its effect on post endodontic pain immediately and after 8,12,24,48 hours after completion of endodontic treatment
  Interventions: Drug: curcumin group:Curcumin is an ancient coloring spice . Interestingly, it has various pharmacological activities including analgesic, anti-inf; Dietary Supplement: 400mg starch
- Starch(400mg starch) starch is sometype of carbohydrates (Placebo Comparator): patints taking(400mg) starch in tabelts in same shape and color of control group before endodontic treatment by one hour and post endodontic pain immediately and after 8,12,24,48 hours after treatment completion
  Interventions: Drug: curcumin group:Curcumin is an ancient coloring spice . Interestingly, it has various pharmacological activities including analgesic, anti-inf; Dietary Supplement: 400mg starch

INTERVENTIONS:
Drug: curcumin group:Curcumin is an ancient coloring spice . Interestingly, it has various pharmacological activities including analgesic, anti-inf — effect of taking 400mg curcumin one hour before endodontic ttt on post endodontic pain immediatelly and after 8,12,24,48 hours after endodontic treatment.Curcumin is an ancient coloring spice of Asia which is powerful antioxidant , it has hepatoprotective effect and traditionally used for many remedies . Interestingly, it has various pharmacological activities including analgesic, anti-inflammatory , It is even reported to have antimicrobial effect .
  Medical clinical trials reported on the analgesic effect of curcuminoids in reducing postsurgical pain osteoarthritis and rheumatoid arthritis .
  other name : curcum, tumeric
  Other Names: curcum-tumeric
Dietary Supplement: 400mg starch — patints taking(400mg) starch in tabelts in same shape and color of control group before endodontic treatment by one hour and post endodontic pain immediately and after 8,12,24,48 hours after treatment completion

SUMMARY:
Will premedication with Curcumin in single endodontic treatment in patients having acute pulpitis in mandibular molars affect post- operative pain?

This the present study hopes to bring an evidence based decision on the possibility of using curcumin as a premedication to reduce post-operative pain in single visit treatment of cases with acute pulpitis

DETAILED DESCRIPTION:
The diagnostic data will be collected in a general health chart and dental history sheet by the investigator and confirmed for eligibility criteria with main supervisor.

Clinical examination through visual, palpation and percussion of offending tooth is done. Pulp sensitivity test will be done for baseline comparison. It will be performed by both by electric and thermal tests on offending tooth and the contralateral. Preoperative periapical radiograph is done to evaluate pulp chamber size and shape, root and root canals and detect any per apical changes.

The selected mandibular molars should have final diagnosis of acute pulpitis.

Diagnostic criteria for acute pulpitis tooth:

Palpation test: not sensitive & Percussion test: not sensitive &Thermal test: hypersensitive to heat or cold & Radiographic: periapical radiograph shows normal periapex • Sequence of procedural steps:

The study protocol is described to the patients and they sign an informed consent . Each patient will be given pain scale chart (VAS) in order to record his /her pain level before any intervention, and then patients will be given the premedication according to the study group:

Group A" intervention or Curcumin group ": (400mg Curcumin) in one capsule Group B" placebo group ": starch capsule, Both capsules of intervention and placebo groups will have the same shape, color and are prepared by Professor Doctor Mohamed Elnabarawy in the faculty of pharmacology, Cairo University. Every patient takes one capsule before endodontic treatment by one hour according to randomization sequence table prepared by the main supervisor utilizing "random.org".

The researcher will give nerve block anesthesia according to the region of the tooth will be treated, ARTINIBSA 4% articaine hydrochloride 4% with 1:100,000 epinephrine as vasoconstrictor will be used.

An access cavity is performed by using round bur and endo-z bur, afterwards. The tooth will be properly isolated with rubber dam. Irrigation is done with 2ml 2.5% Sodium hypochlorite (Clorox, Nobelwax Factories for chemicals, Egypt) , then canal negotiation with K-file #15 (K-file, Dentsply Maillefer , Switzerland), and working length will be determined using an electronic apex locator (iPex NSK,Japan) and confirmed radiographically, sequentionaly larger file sizes will be introduced to the working length to gague the initional apical file size.

Mechanical preparation will be performed by crown-down technique using rotary M-Pro files, in an endodontic motor (Endo mate, NSK, Japan) with adjusted torque and speed according to the manufacturer's instructions ( 450 rpm -1.5 Ncm). Gauging apical diameter will be done with manual files to determine the master apical file size. If necessary; further larger apical preparation will be done with by manual files. The rotary files will be introduced inside the canal lubricated with EDTA Cream (MD-Chelcream, META BIOMED CO, Korea) The canals are thoroughly irrigated using 2.5% NaOCl between every subsequent instrument by using side vented needle, 27 gauge, with maximum depth of working length - 1mm. The irrigant is delivered having 2ml volume at a rate 1ml/30 second.

Root canal is dried using sterile paper points corresponding to master cone size followed by doing master cone periapical radiograph by ViVi, S.r.I, Italy- X-ray machine and intraoral periapical Kodak Dental film, speed D, #2.

Obturation of the canals is done by lateral compaction technique and master cone cementated by resin sealer (ADSEAL, META BIOMED CO., Korea). A spreader #30 will be used 2mm short of working length to allow for auxiliary cones #25, taper 2% to be added and excess will be removed with hot instrument up to cervical line followed by insertion of temporary filling to seal the access cavity.

Post-operative periapical radiograph is taken after obturation. Pain will be assessed by giving the patient the pain scale (VAS) to assess pain immediately after treatment and at 8, 12,24,48 hours after the visit.

VAS pain scale is horizontal scale from1-100mm.patient mark on the scale and investigator will measure with ruler and conert to cateigories as follow (0-40mm): no pain, (5-44mm) : mild, (45-74mm): moderate,(75-100) .

Patients will come back at clinic after 48hours and deliver their signed scoring sheet and referred to restorative department for permanent restoration.

• In case of post appointment emergency cases:

The pain is recorded by pain scale and emergency treatment done according to pain severity; recording of pain scale is continued according to schedule time line. Sequence of emergency treatment includes:

1. Make sure the tooth is out of occlusion
2. Hot saline mouth bath
3. When pain is moderate /severe: Anti- inflammatory: ibuprofen600 tab/8hr (6)
4. Antibiotics (is only prescribed in presence of swelling and/or systemic manifestations as malaise or palpable lymph nodes or fever) Hibiotic 1gm tab/12hrs and Flagel 500 mg tab/12 hrs for 5 days N.B if allergic to penicillin; Dalacin C 300 mg cap/8hrs for 5days

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Patients with age range 20- 55y
* Mandibular molars with acute pulpitis.
* Teeth with mature root

Exclusion Criteria:

* Pregnant or lactating females
* Teeth with non vital pulp
* Non- restorable teeth
* Medically compromised patients(diabetics-bleeding disorder- hypertensive )
* Patients with facial swelling or acute infection.
* Previously endodontically treated teeth
* Periodontally affected teeth.
* Teeth with calcified root canals, root caries, internal or external root resorption, sign of crack formation and anatomic abnormalities.
* Patients taking analgesic medication before 12hours.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
change in post operative pain after single endodontic visit | immediately and after 8,12,24,48 hours after completion endodontic treatment
  intenisty of postoperative pain by using VAS pain scale which is horizontal scale from0-100mm which patient will on degree of his/her pain level and investigator will measure it with ruler and convert to catogries as follow (0-4mm): no pain, (5-44mm) : mild, (45-74mm): moderate,(75-100) : severe.

SECONDARY OUTCOMES:
number of analgesic tablets taken | immediately and after 8,12,24,48 hours after completion endodontic treatment
  counting of analgesic tablets taken from rescue medication (ibuprofen600 tab)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt

REFERENCES:
- [Background] Taylor H, Warfield CA. Thermography of pain: instrumentation and uses. Hosp Pract (Off Ed). 1985 Nov 15;20(11):164, 168-9. doi: 10.1080/21548331.1985.11703194. No abstract available. PMID 2997245
- [Background] Praveen R, Thakur S, Kirthiga M. Comparative Evaluation of Premedication with Ketorolac and Prednisolone on Postendodontic Pain: A Double-blind Randomized Controlled Trial. J Endod. 2017 May;43(5):667-673. doi: 10.1016/j.joen.2016.12.012. Epub 2017 Mar 17. PMID 28320541
- [Background] Arslan H, Topcuoglu HS, Aladag H. Effectiveness of tenoxicam and ibuprofen for pain prevention following endodontic therapy in comparison to placebo: a randomized double-blind clinical trial. J Oral Sci. 2011 Jun;53(2):157-61. doi: 10.2334/josnusd.53.157. PMID 21712619
- [Background] Mokhtari F, Yazdi K, Mahabadi AM, Modaresi SJ, Hamzeheil Z. Effect of Premedication with Indomethacin and Ibuprofen on Postoperative Endodontic Pain: A Clinical Trial. Iran Endod J. 2016 Winter;11(1):57-62. doi: 10.7508/iej.2016.01.011. Epub 2015 Dec 24. PMID 26843879